CLINICAL TRIAL: NCT01842477
Title: Evaluation of Efficacy and Safety of Autologous MSCs Combined to Biomaterials to Enhance Bone Healing in Patients With Delayed Consolidation After Long Bone Fracture Requiring Graft Apposition or Alternative Orthobiologics
Brief Title: Evaluation of Efficacy and Safety of Autologous MSCs Combined to Biomaterials to Enhance Bone Healing
Acronym: OrthoCT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C11-12; 2011-005441-13 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-04-29 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2017-11

CONDITIONS: Delayed Union After Fracture of Humerus, Tibial or Femur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation surgery (Experimental): All the patients will have the implantation surgery. This trial is a one-arm study.
  Interventions: Procedure: Implantation of bone substitute plus autologous cultured mesenchymal cells

INTERVENTIONS:
Procedure: Implantation of bone substitute plus autologous cultured mesenchymal cells — Implantation surgery of a synthetic bone substitute associated with autologous bone marrow cells expanded

SUMMARY:
Bone grafting is widely used in hospitals to repair injured, aged or diseased skeletal tissue. In Europe, about one million patients encounter a surgical bone reconstruction annually and the numbers are increasing due to our ageing population. Bone grafting intends to facilitate bone healing through osteogenesis (i.e. bone generation) at the site of damage, but this is only attained presently by including cells capable of forming bone into the augmentation.

Bone autograft is the safest and most effective grafting procedure, since it contains patient's own bone growing cells (to enhance osteogenesis) and proteins (to enhance osteoinduction), and it providing a scaffold for the new bone to grow into (osteoconduction). However, bone autograft is limited in quantity (about 20 cc) and its harvesting (e.g. from the iliac crest) represents an additional surgical intervention, with frequent consequent pain and complications.

We hypothesize that using autologous bone marrow cells expanded in GMP facility surgically implanted with synthetic bone substitutes contribute to the resolution of the health and socioeconomic complications of delayed union or non-union after diaphyseal and metaphyseal-diaphyseal fractures with safety and efficacy.

DETAILED DESCRIPTION:
Tissue engineering combines bone marrow cells or mesenchymal stem cells (MSCs), synthetic scaffolds and molecular signals (growth or differentiating factors) in order to form hybrids constructs. For bone reconstruction purposes, human MSCs have been seeded and cultured on porous calcium phosphate ceramics in osteogenic media. Some clinical studies with low numbers of patients have been reported using this approach but the outcomes were inconsistent with low efficacy in bone regeneration. The reasons of the limited clinical success may be due to several bottlenecks in the multidisciplinary field of bone tissue engineering. The association in vitro of biomaterials and osteoprogenitor cells raises technical challenges and regulatory and ethic issues for the implementation of clinical trials, whereas the expansion of MSCs is now possible in GMP Facility.

The expected results are to obtain bone consolidation thus healing of delayed union or non-union, as proven by imaging techniques, without using bone graft. This will prove the efficacy of the proposed IMP based on pluripotent MSCs expanded in a GMP facility and mixed with granulated biphasic calcium phosphate in the surgical setting before implantation. No expected complications related to the procedure are expected. Changes in serum levels of bone turnover markers will be described.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65, both sexes
* Traumatic isolated closed or open Gustilo I and II humerus, tibial or femur diaphyseal or metaphyseal-diaphyseal fracture status delayed union or non-union
* At least 3 months from acute fracture
* Able to provide informed consent, and signed informed consent
* Patients (by themselves) should have medical health care coverage to be included in a research study
* Able to understand and accept the study constraints

Exclusion Criteria:

* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control
* Participation in another therapeutic trial in the previous 3 months
* Delayed union or non-union related to iatrogeny
* Segmental bone loss requiring specific therapy (bone transport, large structural allograft, megaprosthesis, etc)
* Vascular or neural injury
* Other fractures causing interference with weight bearing
* Acute persistent chronic bacterial infections such as brucellosis, typhus, leprosy, relapsing fever, melioidosis and tularemia
* Visceral injuries of diseases interfering with callus formation (cranioencephalic trauma, etc.)
* History of bone harvesting on iliac crest contraindicating bone-marrow aspiration
* Corticoid or immunosuppressive therapy more than one week in the three months prior to study inclusion
* History of prior or concurrent diagnosis of HIV-, Syphilis, Hepatitis-B- or Hepatitis-C-infection (confirmed by serology or PCR)
* History of neoplasia or current neoplasia in any organ
* Subject legally protected, under legal guardianship, deprived of their liberty by judicial or administrative decision, subject of psychiatric care, or admission to a health facility.
* Impossibility to meet at the appointments for the follow up
* Insulin dependent diabetes
* Obesity (BMI > 30)
* Autoimmune inflammatory disease
* Current treatment by biphosphonate or stopped in the three months prior to study inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02-05 (Actual); Study Completion 2016-02-05 (Actual)

PRIMARY OUTCOMES:
Complication rate as percentage of patients with local complications regarding the non-union treatment in the follow-up | At 6 weeks, 12 weeks, 24 weeks and 52 weeks after the implantation surgery

SECONDARY OUTCOMES:
Number of patients with proven bone healing | 6 weeks, 12 weeks, and 24 weeks after the implantation surgery
Amount of radiological callus | 6 weeks, 12 weeks, and 24 weeks after the implantation surgery
Clinical consolidation | 6 weeks, 12 weeks, and 24 weeks after implantation surgery
No reoperation done or scheduled | 24 weeks after implantation surgery
Changes in serum levels of bone turnover markers | 6 weeks, 12 weeks, and 24 weeks after the implantation surgery

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gomez Barrena, Principal Investigator — Universidad Autonoma de Madrid
Locations (5):
- France (2):
  - Depatment of Orthopaedic Surgery, Hôpital Henri Mondor, Créteil
  - Department of Orthopaedic Surgery, CHRU Tours, Tours
- Department of Orthopaedic Trauma, University of Ulm, Ulm, Germany
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy
- Servicio de Cirugía Ortopédica y Traumatología "A", Hospital La Paz, Madrid, Spain

REFERENCES:
- [Background] Gomez-Barrena E, Rosset P, Gebhard F, Hernigou P, Baldini N, Rouard H, Sensebe L, Gonzalo-Daganzo RM, Giordano R, Padilla-Eguiluz N, Garcia-Rey E, Cordero-Ampuero J, Rubio-Suarez JC, Stanovici J, Ehrnthaller C, Huber-Lang M, Flouzat-Lachaniette CH, Chevallier N, Donati DM, Ciapetti G, Fleury S, Fernandez MN, Cabrera JR, Avendano-Sola C, Montemurro T, Panaitescu C, Veronesi E, Rojewski MT, Lotfi R, Dominici M, Schrezenmeier H, Layrolle P. Feasibility and safety of treating non-unions in tibia, femur and humerus with autologous, expanded, bone marrow-derived mesenchymal stromal cells associated with biphasic calcium phosphate biomaterials in a multicentric, non-comparative trial. Biomaterials. 2019 Mar;196:100-108. doi: 10.1016/j.biomaterials.2018.03.033. Epub 2018 Mar 19. PMID 29598897
- [Background] Granchi D, Gomez-Barrena E, Rojewski M, Rosset P, Layrolle P, Spazzoli B, Donati DM, Ciapetti G. Changes of Bone Turnover Markers in Long Bone Nonunions Treated with a Regenerative Approach. Stem Cells Int. 2017;2017:3674045. doi: 10.1155/2017/3674045. Epub 2017 Jun 20. PMID 28744314
- See also: Related Info — http://www.reborne.org/